CLINICAL TRIAL: NCT01697748
Title: A Prospective Randomized Study Assessing Post Operative Wound Infections Along With Cosmetic Outcomes Using Silver Impregnated Dressings Compared to Conventional Dressings on Cesarean Section Incisions
Brief Title: Prospective Study on Cesarean Wound Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USF IRB 00008650; NCT01927211 (obsolete NCT alias)
Record Dates: First submitted 2012-09-19; First posted 2012-10-02 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2012-12

CONDITIONS: Surgical Site Infection; Cosmetic Appearance of Cesarean Scar; Post Operative Pain
Keywords: cesarean section incisions; silver; c-section; wound infection; scar appearance; post operative pain
MeSH Terms: conditions — Surgical Wound Infection; Pain, Postoperative; Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telfa pad dressing (Placebo Comparator): Telfa pad dressing placed over Cesarean wound after skin closure; the dressing will be changed to a new Telfa pad dressing on post-operative day 2 which will remain on the incision through post-operative day 7.
  Interventions: Device: Telfa pad dressing
- Silver-impregnated dressing (Active Comparator): Silver-impregnated dressing placed over Cesarean wound after skin closure; the dressing will be changed to saline-treated dressing on post-operative day 2 which will remain on the incision through post-operative day 7.
  Interventions: Device: Silver-impregnated dressing

INTERVENTIONS:
Device: Silver-impregnated dressing — Silver-impregnated dressing placed over Cesarean wound after skin closure; the dressing will be changed to saline-treated dressing on post-operative day 2 which will remain on the incision through post-operative day 7.
  Other Names: Silverlon
  Arms: Silver-impregnated dressing
Device: Telfa pad dressing — Telfa pad dressing placed over Cesarean wound after skin closure; the dressing will be changed to a new Telfa pad dressing on post-operative day 2 which will remain on the incision through post-operative day 7.
  Other Names: Telfa pad
  Arms: Telfa pad dressing

SUMMARY:
This study will investigate whether the placement of silver impregnated dressings beginning in the OR will improve wound healing in patients undergoing cesarean delivery compared to traditional Telfa pads. This study will also explore the presumed improvement in scar integrity when silver impregnated dressings are used compared to the Telfa pads.

The study will compare the percentage of patients who develop a surgical site infection after application of silver impregnated dressings versus standard Telfa dressings. Investigators will also assess the cosmetic appearance and pain of the cesarean section scar at the patient's one week and 6 week post-operative visits.

DETAILED DESCRIPTION:
This is a randomized, prospective study involving 660 patients undergoing cesarean sections at Tampa General Hospital. The control group (n=330) will receive standard Telfa pad dressing and the treatment group (n=330) will receive the silver impregnated dressing.

The primary objective is to compare the percentage of patients who develop a surgical site infection between the two groups at the 1-week and 6-weeks post operative visits. The secondary objective is to assess the cosmetic outcome of the cesarean incision observed at the 1-week and 6-week post-operative visits. A plastic surgery investigator will also conduct a blinded assessment of cosmetic outcome by review of photographs taken of the wounds at 1-week and 6-weeks.The tertiary objective is to evaluate the amount of narcotic and non narcotic medicine consumed during the hospitalization and query the patient with regards to pain involving the cesarean wound at 1 and 6 week post-operative visits

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Elective and emergent cesarean deliveries
* Primary and repeat cesarean sections
* Transverse skin incisions (Pfannenstiel)
* Low transverse uterine incisions
* Patients with or without the diagnosis of chorioamnionitis with antibiotic treatment prior to or after the delivery of the baby
* Single and multiple gestations
* Able and willing to provide written informed consent

Exclusion Criteria:

* Patients that did not receive routine prophylactic dose of antibiotics in the operating room.
* Skin incisions other than Pfannenstiel
* Uterine incisions other than low transverse
* Patients with known or discovered allergy to silver or nylon

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2013-09; Primary Completion 2016-08 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Connery, MD, Principal Investigator — USF Health Morsani College of Medicine, Department of Obstetrics and Gynecology
Locations (3):
- United States (3):
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - Women's Center Operating Rooms at the Tampa General Hospital, Tampa, Florida
  - USF Health Morsani Center for Advanced Healthcare, Tampa, Florida

REFERENCES:
- [Background] Opoien HK, Valbo A, Grinde-Andersen A, Walberg M. Post-cesarean surgical site infections according to CDC standards: rates and risk factors. A prospective cohort study. Acta Obstet Gynecol Scand. 2007;86(9):1097-102. doi: 10.1080/00016340701515225. PMID 17712651
- [Background] Owens SM, Brozanski BS, Meyn LA, Wiesenfeld HC. Antimicrobial prophylaxis for cesarean delivery before skin incision. Obstet Gynecol. 2009 Sep;114(3):573-579. doi: 10.1097/AOG.0b013e3181b490f1. PMID 19701037
- [Background] Olsen MA, Butler AM, Willers DM, Devkota P, Gross GA, Fraser VJ. Risk factors for surgical site infection after low transverse cesarean section. Infect Control Hosp Epidemiol. 2008 Jun;29(6):477-84; discussion 485-6. doi: 10.1086/587810. PMID 18510455
- [Background] Epstein NE. Do silver-impregnated dressings limit infections after lumbar laminectomy with instrumented fusion? Surg Neurol. 2007 Nov;68(5):483-5; discussion 485. doi: 10.1016/j.surneu.2007.05.045. PMID 17961738
- [Background] Perkins James, Pattillo Rolandid. How to Avert Postoperative Wound Complications-Treat It when It Occurs. OBG Management 2009;21(10):43-53.
- [Background] Huckfeldt R, Redmond C, Mikkelson D, Finley PJ, Lowe C, Robertson J. A clinical trial to investigate the effect of silver nylon dressings on mediastinitis rates in postoperative cardiac sternotomy incisions. Ostomy Wound Manage. 2008 Oct;54(10):36-41. PMID 18927482
- [Background] Leaper DJ. Silver dressings: their role in wound management. Int Wound J. 2006 Dec;3(4):282-94. doi: 10.1111/j.1742-481X.2006.00265.x. PMID 17199764
- [Background] Mustoe TA, Cooter RD, Gold MH, Hobbs FD, Ramelet AA, Shakespeare PG, Stella M, Teot L, Wood FM, Ziegler UE; International Advisory Panel on Scar Management. International clinical recommendations on scar management. Plast Reconstr Surg. 2002 Aug;110(2):560-71. doi: 10.1097/00006534-200208000-00031. PMID 12142678
- [Background] Cromi A, Ghezzi F, Gottardi A, Cherubino M, Uccella S, Valdatta L. Cosmetic outcomes of various skin closure methods following cesarean delivery: a randomized trial. Am J Obstet Gynecol. 2010 Jul;203(1):36.e1-8. doi: 10.1016/j.ajog.2010.02.001. Epub 2010 Apr 24. PMID 20417924
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Thomas Steve. MRSA and the Use of Silver Dressings: Overcoming Bacterial Resistance. http://www.worldwidewounds.com/2004/november/Thomas/Introducing-Silver Dressings.html.
- [Background] Yiannias, James. Clinical features and diagnosis of allergic contact dermatitis. http://www.uptodate.com/contents/clinical-features-and-diagnosis-of-allergic-contact-dermatitis
- [Derived] Connery SA, Yankowitz J, Odibo L, Raitano O, Nikolic-Dorschel D, Louis JM. Effect of using silver nylon dressings to prevent superficial surgical site infection after cesarean delivery: a randomized clinical trial. Am J Obstet Gynecol. 2019 Jul;221(1):57.e1-57.e7. doi: 10.1016/j.ajog.2019.02.053. Epub 2019 Mar 5. PMID 30849351

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from September 2013 through June 2016. The 6 week post operative visits were completed August 2016.
  Recruitment was at University of South Florida South Tampa Campus, Tampa General Hospital Healthpark Genesis and Tampa General Hospital Tampa Florida Labor and Delivery Triage.
Pre-assignment Details: 3 patients were inadequately consented, two in the Silverlon dressing group and one in the Telfa dressing group
Period: Overall Study
Arm/Group | Telfa Pad Dressing | Silver-impregnated Dressing
Started | 329 | 328
Completed | 271 | 260
Not Completed | 58 | 68
Not completed — ineligible skin incision | 1 | 2
Not completed — ineligible uterine incision | 4 | 1
Not completed — Lost to Follow-up | 53 | 65

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telfa Pad Dressing | Silver-impregnated Dressing | Total
Number analyzed (Participants) | 329 | 328 | 657
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 329 | 328 | 657
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (5.5) | 30.9 (5.6) | 31.0 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 329 | 328 | 657
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 329 | 328 | 657

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Develop a Surgical Site Infection
Description: A surgical site infection involving the skin and subcutaneous tissue is defined as either
  * The presence of a purulent discharge from the wound on inspection, or
  * Purulent discharge obtained from the wound after exploration based on the suspicion of the provider (erythema, swelling, heat or pain), or
  * The presence of a seroma or hematoma discharge from the wound on inspection or after exploration that also involves isolation of an organism from an aseptically obtained culture based on suspicion of the provider (erythema, swelling, heat or pain). Seromas or hematomas with negative cultures will not be considered a surgical site infection.
Time Frame: from post operative day #1 through post operative day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Telfa Pad Dressing | Silver-impregnated Dressing
Number analyzed (Participants) | 329 | 328
Participants | 14 | 15
Statistical Analysis 1: Comparison: Telfa Pad Dressing vs Silver-impregnated Dressing; With an SSI rate of 15% at Tampa General Hospital at the time of study design, a sample size of 600 patients was determined to provide a power of 80% to detect a 50% absolute reduction (15 vs. 7.5%) surgical site infection at a two sided alpha = 0.05. Assuming an approximate 10% dropout loss to follow up rate, the total sample size was adjusted to 660; Test type: Superiority — With an SSI rate of 15% at Tampa General Hospital at the time of study design, a sample size of 600 patients was determined to provide a power of 80% to detect a 50% absolute reduction (15 vs. 7.5%) surgical site infection at a two sided alpha = 0.05. Assuming an approximate 10% dropout loss to follow up rate, the total sample size was adjusted to 660; Variables with at least a borderline association with a treatment arm (P≤ .10) were included in a multiple logistic regression model to verify which is independently associated with the outcome of interest; No P values were reported for the association between dressing type and infection, only relative risk and 95% confidence intervals were reported; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.44 to 1.96]; Besides the Chi Square, Fisher's Exact test, Student T-test, Mann Whitney U test, and logistic regression were utilized where appropriate
Statistical Analysis 2: Comparison: Telfa Pad Dressing vs Silver-impregnated Dressing; Test type: Superiority — With an SSI rate of 15% at Tampa General Hospital at the time of study design, a sample size of 600 patients was determined to provide a power of 80% to detect a 50% absolute reduction (15% vs. 7.5%) surgical site infection at a two side alpha = 0.05. Assuming an approximate 10% dropout loss to follow up rate, the total sample size was adjusted to 660; p < 0.05, Mixed Models Analysis — Variables with at least a borderline association (P≤.10) were then included in a multiple logistic regression model to verify which is independently associated with the outcome of interest; In addition to the Chi-Square, Fisher's exact test, Student T-Test, Mann Whitney U test and logistic regression were utilized when appropriate

2. Secondary Outcome: Cosmetic Outcome of the Cesarean Section Incision
Description: The following instruments will be used to determine the cosmetic outcome:
  • The Modified Vancouver scar scale Range of scale values are from 0-12 (0 indicating a better outcome)
Time Frame: Post operative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telfa Pad Dressing | Silver-impregnated Dressing
Number analyzed (Participants) | 329 | 328
score on a scale | 3.8 (1.8) | 3.7 (1.8)
Statistical Analysis 1: Comparison: Telfa Pad Dressing vs Silver-impregnated Dressing; Test type: Superiority; p < .05, see below; Chi square, Fisher Exact, Student t-test, Wilcoxon-Mann-Whitney test where appropriate; In addition to Chi-Square, Fisher's Exact test, Student T-test, Wilcoxon-Mann Whitney test were utilized where appropriate

3. Secondary Outcome: Cosmetic Outcome of the Cesarean Section Incision
Description: The following instruments will be used to determine the cosmetic outcome
  • The Modified Observer Scar Assessment Scale Range of scale values is from 5 - 50 ( the lower the score the better the outcome)
Time Frame: Six weeks post-operative
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telfa Pad Dressing | Silver-impregnated Dressing
Number analyzed (Participants) | 329 | 328
score on a scale | 11.4 (6.5) | 11.6 (6.5)
Statistical Analysis 1: Comparison: Telfa Pad Dressing vs Silver-impregnated Dressing; Test type: Superiority; p < .05, Mixed Models Analysis; Chi Square, Fisher's Exact, Student's T test, Wilcoxon-Mann-Whitney test and logistic regression when appropriate,; Besides the Chi Square, Fisher's Exact test, Student T-test, Wilcoxon-Mann-Whitney Test, and logistic regression were utilized where appropriate
Statistical Analysis 2: Comparison: Telfa Pad Dressing vs Silver-impregnated Dressing; Test type: Superiority; p < .05, Mixed Models Analysis; Chi Square, Fisher Exact, Student t-test, Wilcoxon-Mann-Whitney test; Besides the Chi Square, Fisher's Exact test, Student T-test, Wilcoxon-Mann-Whitney test and logistic regression were utilized where appropriate

4. Other Pre Specified Outcome: Reduction of Pain After Cesarean Delivery
Description: The amount of narcotics measured in Morphine equivalent milligrams and non opioids administered during the cesarean delivery hospitalization were recorded
Time Frame: Immediately post operatively to hospital discharge
Measure: Median (Inter-Quartile Range); unit: Morphine milligram equivalent
Arm/Group | Telfa Pad Dressing | Silver-impregnated Dressing
Number analyzed (Participants) | 329 | 328
Morphine milligram equivalent | 90.0 [60 to 135] | 82.5 [52.5 to 120]

5. Other Pre Specified Outcome: The Number of Participants Noting Pain at the One Week Post Cesarean Visit
Description: Pain response to notable pain at wound site during 7 day post operative visit Subjective self reporting pain as yes or no.
Time Frame: Post operative day 7
Population: This was the number of participants that completed the form at their 7 day post- operative visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Telfa Pad Dressing | Silver-impregnated Dressing
Number analyzed (Participants) | 299 | 296
Participants | 23 | 21
Statistical Analysis 1: Comparison: Telfa Pad Dressing vs Silver-impregnated Dressing; Test type: Superiority; p < 0.05, Mixed Models Analysis; [other analysis details as in outcome 3, analysis 1]

6. Other Pre Specified Outcome: The Number of Participants Noting Pain at the Six Weeks Post Cesarean Visit
Description: Pain response to notable pain at wound site during 6 week post operative visit Subjective self reporting of pain as yes or no.
Time Frame: 6 weeks post operative
Measure: Count of Participants; unit: Participants
Arm/Group | Telfa Pad Dressing | Silver-impregnated Dressing
Number analyzed (Participants) | 263 | 242
Participants | 5 | 8
Statistical Analysis 1: Comparison: Telfa Pad Dressing vs Silver-impregnated Dressing; Test type: Superiority; p < 0.05, Mixed Models Analysis; In addition to the Chi-square, Fisher's exact test, Student T-Test, Wilcoxon-Mann-Whitney test and logistic regression were utilized where approprate

ADVERSE EVENTS:
Arm/Group | Telfa Pad Dressing | Silver-impregnated Dressing
All-Cause Mortality (participants affected / at risk) | 0/329 | 0/328
Serious Adverse Events (participants affected / at risk) | 1/329 | 2/328
Other Adverse Events (participants affected / at risk) | 3/329 | 2/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telfa Pad Dressing (N=329) | Silver-impregnated Dressing (N=328)
Readmission to hospital (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telfa Pad Dressing (N=329) | Silver-impregnated Dressing (N=328)
Skin reaction to adhesive (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The application was initiated in 12/12. A sponsor subsequently was identified with the addition of objectives to the study. After completion of the University Clinical Trials agreement by both parties and IRB notification, the clinical trials registration was completed with receipt in 8/13. Patients were then consented and the first randomized patient occurred 9/13.